CLINICAL TRIAL: NCT00415493
Title: Nasal Physiologic Reactivity of Nonallergic Rhinitics to Cold Air Provocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associated Scientists to Help Minimize Allergies (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Stephen A. Tilles MD, Executive Director, Associated Scientists to Help Minimize Allergies
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: AI-005 NAR
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Vasomotor Rhinitis
Keywords: rhinitis; non-allergic rhinitis; rhinomanometry; cold air; triggers: cold, dry air inhalation; warm, most air inhalation; Nonallergic rhinitis; normal controls
MeSH Terms: conditions — Rhinitis, Vasomotor; Rhinitis; Common Cold

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Order 1 (Experimental): Cold-dry air provocation followed (on a separate day) by Warm-moist air provocation
  Interventions: Other: Cold-dry air provocation; Other: Warm-moist air provocation
- Order 2 (Experimental): Warm-moist air provocation followed (on a separate day) by Cold-dry air provocation
  Interventions: Other: Cold-dry air provocation; Other: Warm-moist air provocation

INTERVENTIONS:
Other: Cold-dry air provocation — 15 minute exposure to cold-dry air by nasal mask
Other: Warm-moist air provocation — 15 minute exposure to warm-moist air by nasal mask

SUMMARY:
This study seeks to compare patients with vasomotor rhinitis ("perennial nonallergic rhinitis," "idiopathic rhinitis") with normal controls with respect to their nasal physiologic reactivity to cold air challenge. Ten vasomotor rhinitis (VMR) patients with nasal symptoms triggered predominantly by cold air, four VMR patients with symptoms triggered predominantly by chemicals, and ten nonallergic, non-rhinitic control subjects will be studied.

DETAILED DESCRIPTION:
After initial screening and verification that subjects can cooperate with active posterior rhinomanometry, subjects will be scheduled for two 15-minute exposure sessions with either: cold-dry air, or warm-moist air. Subjects will rate symptoms (and have their nasal airway resistance measured in triplicate) prior to exposure and at 15-min. intervals post-exposure until an hour has passed.

ELIGIBILITY:
Inclusion Criteria:

(cases; n = 14 total; 10 with predominantly "physical" and 4 with predominantly "irritant"triggers):

* A significant history of chronic and/or recurrent nasal symptoms (rhinorrhea, blockage,sneezing or pruritus) in response to:

  1. Changes in temperature and/or humidity predominantly ("physical triggers"; n = 10); or
  2. Two or more nonspecific irritant triggers predominantly, including: perfumes or colognes,cleaning products, environmental tobacco smoke, vehicular exhaust, paint odors, etc. ("irritant triggers";n = 4). This history shall be of at least two years' duration.

Exclusion Criteria:

(controls; n = 10):

* A significant history of chronic and/or recurrent nasal symptoms (rhinorrhea, blockage,sneezing or pruritus) in response to one or more nonallergic triggers, including: perfumes or colognes, cleaning products, environmental tobacco smoke, vehicular exhaust, paint odors, changes in temperature and/or humidity.

Exclusion criteria:

(all subjects; n = 24):

* A prior history of allergic disease (allergic rhinitis, asthma, angioedema, anaphylaxis)
* Significant skin test reactivity to one or more substances in a panel of 24 locally relevant seasonal and perennial aeroallergens
* Negative wheal response to positive control (histamine) on skin test panel
* Abnormalities on a screening x-ray (Waters view) of the paranasal sinuses
* Cigarette smoking (active, within previous 6 months or cumulative history of >20 pack years)
* Chronic cardiopulmonary diseases (asthma, COPD, coronary artery disease…)
* Continuous therapy with medications having antihistaminic or autonomic primary or secondary effects (e.g., oral or topical antihistamines, tricyclic antidepressants, ipratropium bromide, albuterol, alpha- or beta-adrenergic blockers...)
* Unable to provide meaningful tracings on screening rhinomanometry.
* Pregnancy (or planned pregnancy within 6 months); positive urinary HCG at screening visit. Patient is a breast feeding female.
* Upper respiratory infection (common cold or sinusitis) within 2 week of screening.
* Patient has participated in a clinical trial involving an investigational drug within 4 weeks of visit 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Shusterman, MD, MPH, Principal Investigator — University of Washington; Stephen A Tilles,, MD, Study Director — ASTHMA, Inc.
Locations (1):
- ASTHMA, Inc., Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cold-dry Air Followed by Warm-moist Air: To control for possible stimulus-order effects, half of the subjects were evaluated pre- and post-exposure to Cold-dry air followed (on a separate day) by Warm-moist air. Exposures lasted 15 minutes, with a one-hour follow-up period.
- Warm-moist Air Followed by Cold-dry Air: To control for possible stimulus-order effects, half of the subjects were evaluated pre- and post-exposure to Warm-moist air followed (on a separate day) by Cold-dry air. Exposures lasted 15 minutes, with a one-hour follow-up period.
Period: Overall Study
Arm/Group | Cold-dry Air Followed by Warm-moist Air | Warm-moist Air Followed by Cold-dry Air
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cases: non-allergic rhinitis subjects
- Controls: normal subjects
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (10.5) | 32.7 (14.6) | 35.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Net Proportional Change in Nasal Airway Resistance
Description: Net proportional change in nasal airway resistance, pre- to post-exposure, cold air minus warm air day, calculated as a time-weighted average over the 1.0 h post-exposure. At each time point (pre-exposure, immediately post-exposure, and at 15-, 30-, 45- and 60 minutes post-exposure), nasal airway resistance (in Pa/L/sec) was measured in triplicate. The average of each of these measures was taken for each time point. The time-weighted average of these averages was then calculated for the post-exposure time points and compared with the baseline average for that individual on that testing day. The proportional change from baseline on that day was then calculated (unit-less measure). The difference between the pre-to-post change on the cold air day minus the pre-to-post change on the warm air day was then calculated (unit-less measure). The net proportional change corrects for both inter- and intra-individual variability, which in the case of nasal airway resistance is considerable.
Time Frame: One hour
Measure: Mean (Standard Error); unit: proportional change (unit-less)
Arm/Group | Cases | Controls
Number analyzed (Participants) | 14 | 10
proportional change (unit-less) | 0.11 (0.27) | 0.04 (0.16)

ADVERSE EVENTS:
Arm/Group | Cases | Controls
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 0/14 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No